CLINICAL TRIAL: NCT05371522
Title: Neuro-inflammation and Post-infectious Fatigue in Individuals With and Without COVID-19
Acronym: COVFATI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, B.N.M. van Berckel, Professor of Molecular Brain Imaging, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021.0333; 2021-000781-15 (EudraCT Number)
Record Dates: First submitted 2022-05-11; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: long COVID, imaging, (neuro)inflammation
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Intervention Model Description: All individuals included will undergo a [18F]DPA-714 positron emission tomography (PET) scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]DPA-714 (Experimental): All individuals included will undergo a [18F]DPA-714 positron emission tomography (PET) scan, irrespective of the existence of post-COVID-19 complaints.
  Interventions: Radiation: [18F]DPA-714 positron emission tomography (PET) scan

INTERVENTIONS:
Radiation: [18F]DPA-714 positron emission tomography (PET) scan — 60 minute dynamic brain [18F]DPA-714 positron emission tomography (PET) scan followed by a 30 minute static whole body positron emission tomography (PET) scan

SUMMARY:
Neuroinflammation can be an important regulator of long COVID, specifically fatigue and cognitive complaints. There is evidence that peripheral inflammation and neuro-inflammation are involved in fatigue and cognitive complaints, but precise pathophysiological mechanisms and causal relationship with viral infections are still unknown. The primary aim of this study is to quantify neuroinflammation with [18F]DPA-714 (TSPO-binding) PET scans in post-COVID-19 patients with and without post-infectious fatigue and cognitive complaints and relate it to cognitive, psychiatric and post-infectious fatigue symptoms.

DETAILED DESCRIPTION:
In this study we will include 20 post-COVID-19 patients (>3 months after diagnosis or discharge from hospital) (50% with post-infectious fatigue and/or cognitive complaints) and 50% without post-infectious fatigue/cognitive complaints; matched for disease severity). We will also include 10 age/sex-matched healthy controls without history of COVID-19 or severe fatigue/cognitive complaints. RS6971 polymorphism of the TSPO receptor will be determined and low affinity binders will be excluded from this study.

The main study parameter is the measurement of in vivo neuroinflammation with a [18F]DPA-714 90 minutes PET scan, alternately capturing brain (60 minutes) and body (30 minutes) with both continuous on-line and manual arterial blood sampling for full quantification ([18F]DPA-714 volume of distribution). The 30-minutes body scan will be performed to examine whole-body inflammation. Brain MRI will be performed for functional and anatomical information. We will use questionnaires and neuropsychological evaluation to assess chronic fatigue, depressive, anxiety and cognitive symptoms, partially for descriptive purposes.

ELIGIBILITY:
Inclusion Criteria for post-COVID-19 individuals:

* The individual was diagnosed with symptomatic COVID-19, confirmed by a positive PCR for SARS-CoV-2, positive SARS-CoV-2 serology or CO-RADS (COVID-19 Reporting and Data System) 4 or 5 on CT-scan, or antigen quicktest, or had typical symptoms and was part of a household in which another person was tested positive by PCR 2 weeks before or after the first day of illness;
* The individual is 3 months after being diagnosed with COVID-19 or after hospital discharge in case the patient was admitted.
* The individual is in the range 40-60 years of age (to ensure radiation safety)
* The individual has sufficient command of the Dutch language
* Genotyping of rs6971 must show that the individual is a mixed or high affinity binder

Additional Inclusion criteria for patients with post-COVID-19 complaints:

* The patient experiences severe levels of fatigue (≥ 40) on the fatigue subscale of the Checklist Individual Strength [CIS-fatigue]) and/or cognitive complaints (≥ 15) on the concentration subscale of the Checklist Individual Strength [CIS-concentration].The severe fatigue or cognitive complaints started with or increased substantially directly after the onset of symptoms of COVID-19;
* The patient reports physical/social disability (≤ 65 on the Rand36 physical functioning subscale or a score of ≥ 10 on the Work and Social Adjustment Scale [WSAS];

Additional Inclusion criteria for individuals without post-COVID-19 complaints:

* The individual experiences no significant levels of fatigue (< 35 on the fatigue subscale of the Checklist Individual Strength [CIS-fatigue]) or cognitive complaints (<15 on the concentration subscale of the Checklist Individual Strength [CIS-concentration]) and does not subjectively major symptoms of fatigue or cognitive complaints. Based upon average of normal population +1SD.
* The individual reports no physical/social disability (> 65 on the Rand36 physical functioning subscale or a score of < 10 on the Work and Social Adjustment Scale [WSAS]

Inclusion Criteria for Healthy Controls:

* Should be negatively tested for COVID-19 trough PCR, serology, antibodies, or via antigen quicktest
* No evidence for substantial fatigue or cognitive complaints as evidenced by the CIS subscale fatigue (<35) and CIS subscale concentration (<15) and does not subjectively major symptoms of fatigue or cognitive complaints. Based upon average of normal population +1SD
* The individual is in the range 40-60 years of age (to ensure radiation safety)
* The individual has sufficient command of the Dutch language
* Genotyping of rs6971 must show that the individual is a mixed or high affinity binder

Exclusion Criteria:

* Rs6971 shows low affinity binding
* Individuals who are unable to lay still for scanning due to claustrophobia or severe back pain or trypanophobia (fear of needles)
* Gross neurological pathology (strategic or lobar infarcts or stroke or neurotrauma) on MRI or CT that may interfere with the interpretation of the PET scan.
* Have a hemoglobin test (Hb) result of < to 8 in males and < to 7 in females;
* Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Females of childbearing potential must not be pregnant (negative serum β-HCG at the time of screening and negative urine β-HCG within 24 hours prior to injection) or breastfeeding at screening.
* Have donated blood within 6 months prior to the [18F]DPA-714 PET scan day;
* The individual has an already known psychiatric or somatic condition that can explain his/her fatigue or major psychiatric disorder other than somatic-symptom disorder (chronic fatigue) as a main diagnosis. We will also screen for the presence of Post-Traumatic Stress Disorder PTSD as a main diagnosis] (PCL-5) which prevalence may be high in this patient group because of traumatic experiences during the acute phase of COVID-19. We will also screen for the presence of depressive disorder as a main diagnosis. To screen for PTSD and depressive disorder we will use the Diagnostic and Statistical Manual of Mental Disorders version 5 and verbally check if (any) symptoms do not meet the requirements for a PTSS or depression diagnostic/classification;
* Current use of benzodiazepines11brg

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Quantitative neuroinflammation as measured with [18F]DPA-714 positron emission tomography (PET) | 60 minute dynamic brain scan
Whole-body inflammation as measured with [18F]DPA-714 positron emission | 30 minute static whole-body scan

CONTACTS AND LOCATIONS:
Overall Officials: Bart NM van Berckel, Prof., Principal Investigator — Radiology & Nuclear Medicine, Amsterdam Neuroscience, Vrije Universiteit Amsterdam, Amsterdam UMC
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No